CLINICAL TRIAL: NCT02963324
Title: Physiologically-based Pharmacokinetic Modeling of Ivermectin in Healthy Human Volunteers - a Single-center, Open-label Pharmacokinetics Study
Brief Title: Physiologically-based Pharmacokinetic Modeling of Ivermectin in Healthy Human Volunteers
Acronym: IVMPBPK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IVMPBPK
Record Dates: First submitted 2016-11-04; First posted 2016-11-15 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ivermectin (Experimental): Single dose of ivermectin 12 mg (as 4 tablets of Stromectol (R) 3 mg) orally
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin
  Other Names: Stromectol

SUMMARY:
The present study assesses the pharmacokinetic profile of Ivermectin (IVM) in healthy human volunteers and aims to create a physiologically-based pharmacokinetic model. Planned indication is the prevention of malaria transmission.

DETAILED DESCRIPTION:
Ivermectin (IVM) is a broad spectrum antiparasitic drug. Recent research indicates that IVM could potentially be used in malaria vector control.

The present study assesses the pharmacokinetic profile of IVM in healthy human volunteers and aims to create a physiologically-based pharmacokinetic model. This model will be used to characterize enterohepatic circulation, serve as a basis for drug-drug and drug-disease-state interaction studies, and simulations of IVM disposition in different populations, with special regard given to adolescents and children. With this, safety in individual administrations can be increased, and mass drug administration programs, e.g. oral IVM as malaria vector control, be simulated and planned to maximize the share of a population that can be included. Capillary blood concentration profiles will also be determined to assess the amount of IVM delivered to mosquitos in malaria vector control programs. Furthermore, this study will validate dried blood spot analytics of IVM which will allow easier procurement of pharmacokinetics (PK) data in the field.

ELIGIBILITY:
Inclusion criteria

* Age 18-65 years old
* Caucasian male or female volunteers
* Body mass index (BMI) 18-30 kg/m2, weight ≥ 50 kg
* Full mental and legal capacity
* Signed informed consent prior to any study related procedure
* Ability to communicate in German or English, sufficient to comprehend and adhere to study protocol
* Normal physical examination, vital signs, laboratory workup, and electrocardiogram (ECG) (in the opinion of investigator)
* No history or presence of surgical or medical conditions that might interfere with absorption, distribution, metabolism, and / or elimination of study drug, and / or which might increase its toxic effects (in the opinion of investigator)
* No ongoing or recent (one month) participation in another clinical trial
* No loss of blood ≥ 250 ml within the last three months
* No known hypersensitivity to study drug or any of its constituents
* No other conditions or circumstances that might interfere with compliance with study protocol (in the opinion of investigator)

Exclusion criteria

* History or presence of hepatic or biliary disease
* History of gastrointestinal surgery, specifically cholecystectomy
* History or presence of alcohol or drug abuse
* History or presence of neurological or psychiatric comorbidities, including psychological therapy
* Other clinically significant concomitant disease states (e.g., renal disease, cardiovascular disease, etc.)
* Intake of prescribed or over-the-counter medications, herbal preparations, and / or vitamin / dietary supplements
* Clinically relevant history or presence of allergy or asthma (in the opinion of investigator)
* Female volunteers: pregnancy as confirmed by laboratory assessment; breast-feeding
* Known hypersensitivity or allergy to class of drugs or the study product
* Women with intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: female participants of childbearing potential, not using and not willing to continue using two medically reliable methods of contraception for the entire study duration, or who are not using any other method considered sufficiently reliable by the investigator in individual cases, for the duration of the study from screening visit to 30 days after end-of-study-examination.
* Please note that female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of ivermectin in whole blood, plasma, and capillary blood | Intermittent sampling for 72 hours after dosing
Time to maximum concentration (Tmax) of ivermectin in whole blood, plasma, and capillary blood | Intermittent sampling for 72 hours after dosing
Area under the curve (AUC) of ivermectin in whole blood, plasma, and capillary blood | Intermittent sampling for 72 hours after dosing

SECONDARY OUTCOMES:
Occurence of adverse events | For 72 hours after dosing
  adverse events (treatment-emergent and/or leading to premature study drug discontinuation).
Laboratory changes | For 72 hours after dosing
  Change from baseline for clinical laboratory tests at the end of the study.
Changes in electrocardiogram (ECG) | For 72 hours after dosing
  Change from baseline in resting 12-channel electrocardiogram (ECG) at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Krähenbühl, MD PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided